CLINICAL TRIAL: NCT04798521
Title: Oregon HIV/Hepatitis and Opioid Prevention and Engagement (OR-HOPE) Study: Tele-HCV Treatment Trial
Brief Title: TeleHepC Treatment Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Comagine Health (Other); HIV Alliance (Other); Oregon Health Authority (Other)
Responsible Party: Principal Investigator, P. Todd Korthuis, MD, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TeleHepC; UH3DA044831 (NIH)
Record Dates: First submitted 2020-06-03; First posted 2021-03-15 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-HCV Treatment (Experimental): Participants allocated to telemedicine intervention arm are scheduled for treatment assessment by a study clinician. For a majority of participants, this will also be the treatment initiation visit. If additional studies are necessary for routine treatment decision making, peers will assist participants in navigating health system barriers and arrangement of second telemedicine visit.
  Interventions: Other: Tele-HCV
- Community Linkage to Care (Active Comparator): Participants allocated to the community linkage-to-care arm will complete screening, be offered enrollment, and undergo informed consent as in the telemedicine arm. Following study inclusion and enrollment, research staff will refer the participant to a local community health clinic to engage in hepatitis C care and seek treatment.
  Interventions: Other: Community Linkage to Care

INTERVENTIONS:
Other: Tele-HCV — Patients will be prescribed HCV medication treatment for 4 weeks at a time. The study pharmacist will check in with the participant by telephone or telemedicine visit at week 0, week 4, and end of treatment to 1) determine general medication tolerance, 2) assess quality of adherence and 3) dispense medications. Peers will assist participants in keeping telehealth appointments and navigating medication pick up or storage. HCV labs will be repeated at 12 weeks post end of treatment and results will be relayed to the participant in the SVR12 follow up visit with the research assistant, along with follow up surveys. Those successfully achieving SVR12 will be counseled on ongoing harm reduction methods. Those showing persistent HCV viremia at 12 weeks post treatment will be referred to community-based HCV treatment providers for treatment re-initiation.
  Arms: Tele-HCV Treatment
Other: Community Linkage to Care — Following study inclusion and enrollment, research staff will refer the participant to a local community health clinic to engage in hepatitis C care and seek treatment. Peers will assist patients to engage with local primary care and health plan resources and will receive an information sheet on optional clinics to attend and questions to ask their provider.
  Arms: Community Linkage to Care

SUMMARY:
The main goal of this study is to test the efficacy of a peer-facilitated telemedicine HCV treatment implementation strategy for people who use drugs versus local HCV treatment referral for achieving HCV sustained viral response at 12 weeks post-treatment (SVR12).

DETAILED DESCRIPTION:
Non-blinded, randomized controlled trial. In-depth qualitative interviews assess attitudes and barriers to treatment.

In Phase 1, potential participants will be pulled from a convenience sample at a Portland clinic providing care for the urban area. An initial target sample of 100 Hepatitis C positive participants will be enrolled for DBS validation. Power will be reassessed based on feedback from receiver operating curve model and additional participants enrolled up to a total of 100 Hepatitis C Positive participants, if necessary. A total of 500 potential participants can be screened expecting 1 in every 4 participants will be positive HCV.

In Phase 2, rural peer care coordinators (PCCs) and research assistants recruit up to 200 PWUD participants from high-needs rural Oregon counties. Study staff specifically target untreated populations recruited from local syringe exchange programs and direct community outreach (e.g. community barbeques, parks, homeless shelters, food pantries, etc.). Participants are encouraged to refer others for study screening.

A subset of up to 40 study participants will complete in-depth qualitative interviews regarding their experiences of hepatitis C treatment.

ELIGIBILITY:
Inclusion Criteria:

1. live in the study area
2. have injected drugs or report recreational opioid use without injection in the last 90 days
3. are age 18 or greater
4. have chronic active, untreated hepatitis C (defined as positive HCV RNA)
5. are seeking treatment for hepatitis C infection.
6. are able to communicate in English (this is due to the fact that less than 5% of the population in which we are targeting will be non-English speaking; see "Non-English Speaking Subjects" for additional information).
7. are enrolled in health insurance

Exclusion Criteria:

1. Have decompensated cirrhosis, defined as Child-Turcotte-Pugh (CTP) score of 7 or greater, or CTP B cirrhosis. CTP scoring is a composite of laboratory metrics (bilirubin, albumin, PT/INR) and clinical findings, including:

   1. increased abdominal or lower extremity swelling
   2. confusion consistent with hepatic encephalopathy
2. Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Central City Concern, Portland, Oregon
  - Comagine Health, Portland, Oregon
  - HIV Alliance, Roseburg, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herink MC, Spencer HC, Cook RR, Gregoire D, Seaman A, Leichtling G, Babiarz J, Korthuis PT. Peer-assisted telemedicine for hepatitis C intervention in people experiencing housing instability. Harm Reduct J. 2026 Feb 5. doi: 10.1186/s12954-026-01408-y. Online ahead of print. PMID 41645194
- [Derived] Seaman A, Cook R, Leichtling G, Herink MC, Gailey T, Cooper J, Spencer HC, Babiarz J, Fox C, Thomas A, Leahy JM, Larsen JE, Korthuis PT. Peer-Assisted Telemedicine for Hepatitis C in People Who Use Drugs: A Randomized Controlled Trial. Clin Infect Dis. 2025 Mar 17;80(3):501-508. doi: 10.1093/cid/ciae520. PMID 39602441
- [Derived] Herink MC, Seaman A, Leichtling G, Larsen JE, Gailey T, Cook R, Thomas A, Korthuis PT. A randomized controlled trial for a peer-facilitated telemedicine hepatitis c treatment intervention for people who use drugs in rural communities: study protocol for the "peer tele-HCV" study. Addict Sci Clin Pract. 2023 May 27;18(1):35. doi: 10.1186/s13722-023-00384-z. PMID 37245041

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tele-HCV Treatment | Community Linkage to Care
Started | 100 | 103
Completed | 63 | 16
Not Completed | 37 | 87

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tele-HCV Treatment | Community Linkage to Care | Total
Number analyzed (Participants) | 100 | 103 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (11.5) | 42.2 (11.0) | 41.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 35 | 77
  Male | 58 | 68 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 96 | 96 | 192
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 9 | 14
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 89 | 90 | 179
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 103 | 203

OUTCOME MEASURES:

1. Primary Outcome: Viral Response
Description: Number of participants with sustained viral response post HCV treatment. The viral response will be measured via a blood test.
Time Frame: 12 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-HCV Treatment | Community Linkage to Care
Number analyzed (Participants) | 63 | 16
Participants | 63 | 16

2. Secondary Outcome: Treatment Initiation
Description: Number of participants who initiated Hepatitis-C Virus (HCV)treatment at 4 weeks post study enrollment.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-HCV Treatment | Community Linkage to Care
Number analyzed (Participants) | 100 | 103
Participants | 85 | 13

3. Secondary Outcome: Treatment Completion
Description: HCV treatment completion, filled final prescription. 90% of HCV pills taken
Time Frame: 36 weeks post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-HCV Treatment | Community Linkage to Care
Number analyzed (Participants) | 100 | 103
Participants | 46 | 9

4. Secondary Outcome: Engagement in Harm Reduction Resources
Description: Participants complete surveys to assess whether or not they are regularly engaging in substance use and harm reduction resources in the community. Surveys conducted a Baseline, 12 weeks, and 36 weeks.
Time Frame: Baseline, 12 weeks, and 36 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-HCV Treatment | Community Linkage to Care
Number analyzed (Participants) | 100 | 103
Participants
  Baseline | 100 | 103
  12 Weeks | 88 | 83
  36 Weeks | 61 | 68

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 1 year a participant was enrolled in the study.
Arm/Group | Tele-HCV Treatment | Community Linkage to Care
All-Cause Mortality (participants affected / at risk) | 3/100 | 2/103
Serious Adverse Events (participants affected / at risk) | 1/100 | 4/103
Other Adverse Events (participants affected / at risk) | 2/100 | 2/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tele-HCV Treatment (N=100) | Community Linkage to Care (N=103)
Cardiac event (Cardiac disorders) | 0 | 1
Gastrointestinal event (Gastrointestinal disorders) | 1 | 0
AIDS-related event (Immune system disorders) | 0 | 1
Overdose, non-fatal (Social circumstances) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tele-HCV Treatment (N=100) | Community Linkage to Care (N=103)
Unintentional injury (Injury, poisoning and procedural complications) | 0 | 1
Psychological event (Psychiatric disorders) | 1 | 1
Gastrointestinal event (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT04798521/Prot_SAP_000.pdf